CLINICAL TRIAL: NCT02469103
Title: The Utility of Second Generation Colon Capsule Endoscopy in Ulcerative Colitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Siew Chien NG, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UC-C2
Record Dates: First submitted 2015-06-09; First posted 2015-06-11 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Colitis, Ulcerative
Keywords: capsule colonoscopy; ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- C2 & colonoscopy (Experimental): C2 and colonoscopy
  Interventions: Device: C2; Procedure: colonoscopy

INTERVENTIONS:
Device: C2 — C2 and colonoscopy will be performed one after another on the same day
Procedure: colonoscopy

SUMMARY:
The purpose of this study is to investigate the accuracy of second generation colon capsule (C2) in evaluating colonic mucosal inflammation of ulcerative colitis patients, using conventional endoscopy as the gold standard.

DETAILED DESCRIPTION:
Consecutive patients with ulcerative colitis will be recruited. Second generation colon capsule endoscopy (C2) and conventional colonoscopy will be performed one after another on the same day. Colonic mucosal inflammation will be scaled by physicians who review C2 videos and those who perform conventional colonosocpies independently. Physicians who review C2 videos and colonoscopists will be blinded to the findings of colonoscopies and C2 videos, respectively.The accuracy of C2 in evaluating mucosal inflammation will be evaluated, using conventional endoscopy as the gold standard.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80 years
* suspected or known UC
* written informed consent

Exclusion Criteria:

* patients with severe UC according to Truelove and Witts' criteria
* current pregnancy/lactating
* patients with a pacemaker or other implanted electromedical device
* the presence of dysphagia
* patients at higher risk of capsule retention (including Crohn's disease, small bowel tumor, radiation enteropathy, previous intestinal surgery, acute abdominal pain without regular defecation)
* patients with a contraindication to bowel preparation (congestive heart failure, renal insufficiency, a life-threatening condition)
* patients with an allergy to polyethylene glycol, sodium phosphate solution, metoclopramide or bisacodyl suppository

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with extent and severity of colonic inflammation | 1 day
  extent and severity of mucosal inflammation will be assessed by each investigation

CONTACTS AND LOCATIONS:
Overall Officials: Siew Ng, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shi HY, Chan FKL, Higashimori A, Kyaw M, Ching JYL, Chan HCH, Chan JCH, Chan AWH, Lam KLY, Tang RSY, Wu JCY, Sung JJY, Ng SC. A prospective study on second-generation colon capsule endoscopy to detect mucosal lesions and disease activity in ulcerative colitis (with video). Gastrointest Endosc. 2017 Dec;86(6):1139-1146.e6. doi: 10.1016/j.gie.2017.07.007. Epub 2017 Jul 14. PMID 28713062